CLINICAL TRIAL: NCT01035424
Title: Genotype-Phenotype Correlations of Late Infantile Neuronal Ceroid Lipofuscinosis
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0901010186; U54NS065768 (NIH); R01NS061848 (NIH); 5R01NS061848-04 (NIH); LDN 6716 (Other: RDCRN)
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Batten Disease; Late Infantile Neuronal Ceroid Lipofuscinosis
Keywords: Batten Disease; Late Infantile Neuronal Lipofuscinosis; LINCL
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to assess the genotype - phenotype correlations of the CNS manifestations of late infantile neuronal ceroid lipofuscinosis (LINCL), a fatal, rare, recessive disorder of the CNS in children. This study will be accomplished by comparing the genotype to a neurologic assessment and Weill Cornell LINCL scale, the UBDRS scale, the standardized CHQ quality of life scale, and the Mullen scale; magnetic resonance imaging (MRI); and routine clinical evaluations. This study is designed to run parallel to a separate study which is being done by the Department of Genetic Medicine, which will use gene transfer to treat the central nervous system (CNS) manifestations of late infantile neuronal ceroid lipofuscinosis.

DETAILED DESCRIPTION:
This protocol is designed to study the natural disease process of LINCL. We propose to assess the correlation between genotype (genetic constitution) and phenotype (observable characteristics) of late infantile neuronal ceroid lipofuscinosis (LINCL) in children diagnosed with LINCL in all stages. LINCL is a form of Batten disease that affects the brain of children and prevents it from functioning properly. These children are born with genetic changes called mutations that result in the inability of the brain to properly recycle proteins in the brain. The recycling failure leads to death of the nerve cells in the brain and progressive loss of brain function. Children with Batten disease are normal at birth but by age 2 to 4 have motor and vision problems which progress rapidly to death at age approximately 10 years old. There are no therapies available to treat the disease. This study is designed to run parallel to the gene transfer protocol, which will include 16 individuals in two groups: Group A will receive 9.0x10^11 genome copies (gc) of the vector and Group B will receive 2.85x10^11 gc; we anticipate that we will be able to capture a one-time genotype - phenotype snapshot for all n=32, and an 18 months genotype - phenotype progression assessment for n=16.

ELIGIBILITY:
Inclusion Criteria.

1. Definitive diagnosis of LINCL, based on clinical phenotype and genotype.
2. The subject must be between the age of 2 and 18 years.
3. The subject will not previously have participated in a gene transfer or stem cell study.
4. Parents of study participants must agree to comply in good faith with the conditions of the study, including attending all of the required baseline and follow-up assessments, and both parents or legal guardians must give consent for their child's participation.

Exclusion criteria.

1. Presence of other significant medical or neurological conditions may disqualify the subject from participation in this study e.g.,malignancy, congenital heart disease, liver or renal failure.
2. Subjects without adequate control of seizures.
3. Subjects with heart disease that would be a risk for anesthesia or a history of major risk factors for hemorrhage.
4. Subjects who cannot participate in MRI studies.
5. Concurrent participation in any other FDA approved Investigational New Drug.
6. Subjects with history of prolonged bleeding or abnormal platelet function or taking aspirin.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be carried out in children diagnosed with LINCL in all stages.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Weill-Cornell LINCL scale at 18 months | Day 0, 18 months
  The Weill Cornell LINCL scale, a 12 point scale which combines assessment of feeding, gait, motor and language to give an overall assessment of various CNS functions
Change in MRI parameters at 18 months | Day 0, 18 months
  MRI assessment at various intervals Day 0 and month 18. Based on previous analyses, we have determined that 3 imaging parameters (% grey matter volume, % ventricular volume and cortical apparent diffusion coefficient) correlate best with age and with the Weill Cornell LINCL scale. These 3 imaging parameters will be used to assess disease progression in this screening protocol and the effect of the gene transfer in the IRB approved gene transfer trials (IRB #0810010013 and #1005011054). For those children available to continue in the study, all parameters will be re-assessed by comparing baseline evaluations to month 18 evaluation.

SECONDARY OUTCOMES:
Change in CHQ or ITQoL | Day 0, 18 months
  Quality of life questionnaires which will be completed by at least one parent/legal guardian at the time of the LINCL patients' visits to Weill Cornell16,17; we will administer either survey depending on the age of the subject independently to each parent to minimize observer bias if both parents are present.
Change in Mullen Scale | Day 0, 18 months
  A pediatric developmental psychological rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No